CLINICAL TRIAL: NCT07152847
Title: Developing a Psychosexual Education App With Artificial Intelligence for National Health Service Patients on a Psychosexual Services Waiting List: A Pilot Pre Test Post Test Study
Brief Title: Developing a Psychosexual Education App With Artificial Intelligence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Metropolitan University (Other)
Collaborators: Homerton University Hospital NHS Foundation Trust (Other); Barts & The London NHS Trust (Other)
Responsible Party: Principal Investigator, Samantha Banbury, Principal Investigator, London Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: T2- SSSP-2025-16
Record Dates: First submitted 2025-09-02; First posted 2025-09-03 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Sexual Dysfunction
Keywords: Psychosexual app; Artificial intelligence; Cognitive mindfulness; Well being; Quality of life
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Artificial Intelligence

STUDY DESIGN:
Intervention Model Description: A pre test post test study will be used to ensure that all participants receive this intervention after providing consent. No control group will be used as the investigators determined that it would be unfair to exclude participants from accessing the app resources. Quality of life and well being will be prioritised, hence the decision to conduct a pre test post test study. Since this is quasi experimental, associations between the app intervention and variable outcomes will be made. Recruitment will be via the National Health Service, for which a separate ethics submission will be made. Recruitment will be based on psychosexual services at the National Health Service. The average waiting list for psychosexual National Health Service services is 6 months. This consideration was necessary when determining the design of this study. There must be no overlap between using the intervention and receiving psychosexual counselling, as this might skew outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre test post test (Other): Repeated measures within subject design
  Interventions: Other: Psychosexual education app with artificial intelligence

INTERVENTIONS:
Other: Psychosexual education app with artificial intelligence — Development of the App will contain the following features:
  1. A basic Mac for iphone Operating System development
  2. General Data Protection Regulation compliance legal certification
  3. Hosting and cloud services
  4. Security Features: for encryption and secure authentication user sign in
  5. Analytics Integration: for integrating app analytics tools
  6. Push Notifications: incorporated into the app
  7. Legal and Compliance additional General Data Protection Regulation certified
  8. Custom Artificial Intelligence Models Interactive Learning Tools Artificial Intelligence will create interactive educational materials on sexual function and dysfunction
  9. Artificial Intelligence cloud services
  10. Natural Language Processing. Artificial Intelligence will process textual data from the feedback questions to identify emerging topics and concerns in sexual function and participants' experiences using the app.

SUMMARY:
The goal of this clinical trial is to establish the effectiveness of a resource based educational psychosexual app for patients attending a waiting list for psychosexual therapy. The app will provide information on sexual dysfunction, kegel exercises, cognitive and mindfulness exercises, along with suitable resources providing information on sexual functioning for men and women. The app will integrate artificial intelligence to improve user experience and efficiency.

The current waiting lists for the National Health Service Psychosexual services are approximately 6 months. Based on this, a pre test post test study measuring participants' sexual functioning, well being, cognitive mindfulness and quality of life will be taken at points 0, 8 and 16 weeks.

Outcomes will assess whether the app was sufficient for these domains. This might further reduce the strain on the National Health Service's resources.

It is hypothesised that app use from weeks 0, 8, and 16 follow up will improve sexual functioning, well being, quality of life, and cognitive mindfulness.

DETAILED DESCRIPTION:
Sexual dysfunction is a group of disorders which affect male and female sexual functioning and negatively impact self-esteem, sexual self efficacy and well being. For women, sexual dysfunction may include sexual interest and arousal disorder, orgasmic disorder, Genito-pelvic pain penetration disorder and substance and medication induced sexual dysfunction. For men, sexual dysfunction may include erectile dysfunction, premature ejaculation or rapid ejaculation, delayed ejaculation, hypoactive sexual desire disorder and substance and medication induced sexual dysfunction.

As part of psychosexual counselling, varied integrative approaches are used quite often, including brief cognitive behavioural therapy, which extends over 6 to 8 sessions. Interventions might also include the use of mindful compassion for varying psychosexual presentations, which are practised in some National Health Services.

An additional adjunct intervention might include psychosexual education. Psychosexual education is diverse and provides information and resources on all aspects of sexual functioning, guidelines and motivational strategies for engaging in varied sexual activities, sexual intimacy and anatomy. Psychosexual education may provide information on sexual health knowledge. These can be delivered in various formats, such as educational programs, face to face education, and internet based and virtual interventions. Recent applications have centred on e learning, including computer based, online and offline presentations. Using an e learning delivery in healthcare services challenges the barriers of resources, time and space. Talking about sex might prove discomforting or embarrassing; for some, cultural, gender or religious factors might further compound open dialogue on sexual matters. Using an e learning approach might target a wider geographic demographic, making it easier for diverse people to access evidence based information whilst minimising discomfort or embarrassment.

One such e learning delivery system is smartphone applications. Most apps included Kegel exercises and working with thoughts and emotions.

Artificial Intelligence has recently been incorporated into apps to improve user experience and efficiency. Artificial intelligence can identify trends in sexual health, behaviour, and attitude. Artificial Intelligence can teach sexuality, sexual health, and behaviour with limited or no human interaction needed.

Limited evidence based psychosexual educational apps are incorporating artificial intelligence to support sexual functioning among men and women. More so among those on a waitlist for National Health Service psychosexual therapeutic support. Indeed, despite the diverse range of biopsychosocial approaches provided by the National Health Service to support sexual dysfunction, waiting lists can be up to 6 months. Therefore, a waiting period without support might further impact sexual function, sexual health, well being and quality of life.

This initial study will target patients on the National Health Service waiting list for psychosexual therapy. This will consist of a psychosexual education app integrating artificial intelligence. Pre test post test measurements will be taken at 0, 8, and 16 weeks, aligning with National Health Service waiting periods. Outcomes will assess well being, quality of life, cognitive mindfulness, sexual functioning, and whether the app was sufficient for participants difficulties. This might further reduce the strain on National Health Service resources.

It is hypothesised that app use from weeks 0, 8, and 16 follow up will improve sexual functioning, well being, quality of life, and cognitive mindfulness.

ELIGIBILITY:
Inclusion Criteria:

* Must be aged 18 years and above
* Must have a laptop, computer, or mobile phone. The App can only be accessed on smartphones and laptops.
* Must have been referred to the National Health Service with a psychosexual presentation
* Must be currently awaiting psychosexual therapy
* Must have been on a National Health Service psychosexual waiting list for less than one month
* Must be fluent in reading and writing English, as this is a clinical trial, the investigators wanted to ensure that participants fully understand what was expected.
* The Patient Health Questionnaire 2 screening for depression must have a score range between 0 to 2 negative
* The Generalised Anxiety Disorder questionnaire 2 screening for anxiety must have a score range between 0 to 2 negative

Exclusion Criteria:

* Aged below 18 years
* Do not possess a mobile phone, computer or laptop
* Are not part of a National Health Service referral system
* Do not have a psychosexual presentation
* Are currently or starting psychosexual therapy
* Have difficulties understanding or speaking English
* The Patient Health Questionnaire 2 screening outcomes 3 and above
* The Generalised Anxiety Disorder questionnaire 2 screening outcomes 3 and above

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self defined male or female based on the assessments used
Enrollment: 150 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Index | 0, 8 and 16 weeks
  This is a 19 item questionnaire on sexual function, including sexual desire, orgasm, lubrication, sexual satisfaction and pain. It has five response categories. Scores include severe 2-7.2, moderate 7.3-14.4, mild to moderate 14.5-21.6, mild 21.7- 28.1 cut-off value, and no female sexual dysfunction 28.2 -36.The lower the score, the higher the level of sexual dysfunction. Cronbach alpha is 0.820 and higher.
The International Index of Erectile Function | 0, 8 and 16 weeks
  This is a 16 item questionnaire on sexual function, including sexual attempts, completed attempts and satisfaction. It has varied response categories. There is a 6 response category for questions 1 to 9 based on sexual attempts. Questions 10 to 15 consist of five response categories, examining sexual satisfaction. Higher scores equate to higher levels of sexual functioning. Cronbach alpha is between 0.80 and 0.90.
Premature Ejaculation Diagnostic Tool | 0, 8 and 16 weeks
  This consists of 5 questions and 3 sections. The first section and question concern delayed ejaculation. For this question, there are five response categories. This is followed by section 2, which consists of two questions based on ejaculation quality and the levels of stimulation required. The third section consists of two questions which address levels of frustration based on a 5 response categories. The higher the score the higher the level of ejaculatory difficulties. The Cronbach alpha is 0.70.

SECONDARY OUTCOMES:
Cognitive mindfulness | 0, 8 and 16 weeks
  This is a 10 item questionnaire with 5 response categories 1 never or rarely true through 5 very often always true. Cronbach's alpha ranges between 0.69 and 0.76. Subscale scoring is divided into five areas: observing, describing, acting with awareness, non judging, and non reactivity. Higher scores indicate greater endorsement of mindfulness.
Short Warwick Edinburgh Mental Wellbeing Scale | 0, 8 and 16 weeks
  A 7 item questionnaire with 5 response categories looking at functioning and feeling aspects of wellbeing. The response categories include 1, none of the time, to 5, all of the time. There is no reverse scoring. Scores range from 7 to 35 where the latter is the highest level of wellbeing. The Cronbach alpha is equal to or greater than 0.70.
Adapted Quality of life questionnaire | 0, 8 and 16 weeks
  This is a 9 item questionnaire with 5 response categories, including 1= strongly agree to 5= strongly disagree, that looks at general, social, and health related quality of life. The higher the score, the higher the quality of life. The Cronbach alpha ranges between 0.70 and 0.90.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Banbury, Principal Investigator — London Met Uni

IPD SHARING:
Plan to Share IPD: No
The National Health Service will anonymise data before analysis. This will need to be confirmed whether the data can be made available for analysis due to ethical considerations.

REFERENCES:
- [Background] Fischer OJ, Marguerie M, Brotto LA. Sexual Function, Quality of Life, and Experiences of Women with Ovarian Cancer: A Mixed-Methods Study. Sex Med. 2019 Dec;7(4):530-539. doi: 10.1016/j.esxm.2019.07.005. Epub 2019 Sep 7. PMID 31501030
- [Background] Dubinskaya A, Heard JR, Choi E, Cohen T, Anger J, Eilber K, Scott V. Female sexual health digital resources: women and health care providers need more options. Sex Med Rev. 2023 Jun 27;11(3):174-178. doi: 10.1093/sxmrev/qead016. PMID 37102305
- [Background] Faubion SS, Rullo JE. Sexual Dysfunction in Women: A Practical Approach. Am Fam Physician. 2015 Aug 15;92(4):281-8. PMID 26280233
- [Background] Jurin T, Sostaric M, Jokic-Begic N, Lauri Korajlija A. mSexHealth: An Overview of Mobile Sexual Health Applications. J Sex Marital Ther. 2023;49(2):129-140. doi: 10.1080/0092623X.2022.2079576. Epub 2022 Jun 2. PMID 35652779
- [Background] Karim H, Choobineh H, Kheradbin N, Ravandi MH, Naserpor A, Safdari R. Mobile health applications for improving the sexual health outcomes among adults with chronic diseases: A systematic review. Digit Health. 2020 Feb 20;6:2055207620906956. doi: 10.1177/2055207620906956. eCollection 2020 Jan-Dec. PMID 32128234
- [Background] Lou IX, Chen J, Ali K, Chen Q. Relationship Between Hypertension, Antihypertensive Drugs and Sexual Dysfunction in Men and Women: A Literature Review. Vasc Health Risk Manag. 2023 Nov 3;19:691-705. doi: 10.2147/VHRM.S439334. eCollection 2023. PMID 37941540
- [Background] Nicol A, Chung E. Male sexual dysfunction: Clinical diagnosis and management strategies for common sexual problems. Aust J Gen Pract. 2023 Jan-Feb;52(1-2):41-45. doi: 10.31128/AJGP-09-22-6559. PMID 36796767
- [Background] Pettigrew JA, Novick AM. Hypoactive Sexual Desire Disorder in Women: Physiology, Assessment, Diagnosis, and Treatment. J Midwifery Womens Health. 2021 Nov;66(6):740-748. doi: 10.1111/jmwh.13283. Epub 2021 Sep 12. PMID 34510696
- [Background] Vosoughi N, Maasoumi R, Haeri Mehrizi AA, Ghanbari Z. The Effect of Psychosexual Education on Promoting Sexual Function, Genital Self-Image, and Sexual Distress among Women with Rokitansky Syndrome: A Randomized Controlled Clinical Trial. J Pediatr Adolesc Gynecol. 2022 Feb;35(1):73-81. doi: 10.1016/j.jpag.2021.06.008. Epub 2021 Jul 13. PMID 34271197